CLINICAL TRIAL: NCT06621290
Title: Understanding the Patient Experience of Geriatric Assessment in the Emergency Department
Brief Title: Patient Experience of CFS-assessment in the ED
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Daniel Wilhelms, MD PhD, University Hospital, Linkoeping
Other Study IDs: 2024-03729-01
Record Dates: First submitted 2024-09-19; First posted 2024-10-01 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Frailty in Aging; Emergency Department Visit; Patient Experience; Qualitative Research

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients over the age of 65 visiting the ED: Patients over the age of 65 visiting the ED who is capable of giving informed consent and who are planned to participate in a frailty assessment
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Semi-structured interviews — Semi-structured interviews on ED-patients experiences of frailty assessment with the CFS
  Other Names: Qualitative research

SUMMARY:
An increasingly common subject of interest among emergency care research is frailty, which is commonly described as a decline in several inter-related physiological systems, in addition to an increased vulnerability to stressors. To increase emergency care staffs ability to intervene appropriately in patients who need interventions to improve their outcomes, geriatric emergency care guidelines include recommendations to identify frailty during the emergency department (ED) visit. However, the patients´ experience of frailty assessment in general is sparsely investigated, and such studies within the ED context are even more limited.

It is conceivable that the patients experience of a frailty assessment may differ depending on several different factors, including which assessment tool is used.

A large number of assessment tools have been developed to help identify frailty, of which the Clinical Frailty Scale (CFS) is one of the most widely used. The CFS has been validated for persons ≥65 years of age and has been evaluated for validity, reliability and feasibility in an ED-setting. The CFS consists of pictograms combined with clinical descriptions of a persons level of functioning in daily life and cognitive status. Hence, to determine the CFS-score, the healthcare staff needs to ask the patient about their physical activity and function level regarding instrumental and personal activities of daily living (eg, banking, shopping, medication management, housekeeping, dressing and hygiene matters).

Since the different questions are often not directly linked to the patients acute illness, but touch on personal subjects like the persons abilities and life situation, it is desirable to understand the patients experience of such an assessment in order to optimise the approach from a patient perspective. To the best of our knowledge, there are no studies that focus on how patients experience being assessed with CFS during their ED-visit.

The aim of this study is therefore to inform a model to guide emergency department staff in assessing frailty with CFS, directed by the perspective from patients along the frailty trajectory. Specifically, our question is:

- How do older ED-patients experience the frailty assessment with the CFS?

DETAILED DESCRIPTION:
With the nature of qualitative data, a definitive sample size cannot be determined in advance. An estimate is that data will need to be collected for 15-25 patients. The analysis is planned to start in parallel with the data collection, and when no further significant findings are made during the progress of the analysis, the data collection will end. To ensure study quality, a reflexive approach and data-/researcher triangulation will be applyed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 65 years attending the ED, and who gives informed consent to participating in the study.
* Emergency department staff will be included if they are to perform a CFS assessment on a patient eligible for the study.

Exclusion Criteria:

* Patients who lack cognitive capacity to give informed consent, or have an acute medical condition will be excluded from the study. Exclusion will also apply to patients who do not speak Swedish and where an interpreter cannot be arranged (the patients next of kin will not be used as an interpreter).
* Exclusion criteria for staff will be unwillingness to give informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over the age of 65, and staff in the ED
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
The patient experience of participating in a frailty assessment with the CFS | immediately after the CFS-assessment
  Qualitative method, conducted in the form of video recordings of the CFS-assessments and individual semi-structured interviews. The planned method of analysis is Thematic Analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Wilhelms, PhD, MD, Principal Investigator — Department of Emergency Medicine in Linköping, and Department of Biomedical and Clinical Sciences, Linköping University, Linköping, Sweden
Locations (1):
- Department of emergency medicine, Linköping University Hospital, Region Östergötland, Linköping, Linköping, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Pseudonymized data may be shared upon request